CLINICAL TRIAL: NCT03702647
Title: Ropivacaine For Post-POEM Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence Charles Hookey (Other)
Responsible Party: Sponsor-Investigator, Lawrence Charles Hookey, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DMED -2186-18
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Achalasia; Esophageal Achalasia
Keywords: Peroral Endoscopic Myotomy; Ropivacaine; Post-procedure pain control
MeSH Terms: conditions — Esophageal Achalasia | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study will be randomized to receive either 30mL of normal saline (placebo), or 30mL of 0.2% ropivacaine in the POEM tunnel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized by an independent research pharmacist to receive either 30mL 0.2% ropivacaine or 30mL of placebo (saline), both being clear, colorless solutions. These samples will be prepared by the research pharmacist 2-3 weeks prior to the procedure and stored until the procedure date as per pharmacy standards. On the morning of the procedure, the study solution will be taken to the operating room with the patient. During the POEM procedure, prior to closure of the mucosotomy, the study solution is instilled into the tunnel. The investigator, patient, care provider, and research coordinator will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Experimental): 30mL of 0.2% Ropivacaine placed in the POEM tunnel
  Interventions: Drug: Ropivacaine
- Normal Saline (Placebo Comparator): 30mL of normal saline placed in the POEM tunnel
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine — 30mL of 0.2% Ropivacaine placed in the POEM tunnel
  Arms: Ropivacaine
Drug: Normal saline — 30mL of normal saline placed in the POEM tunnel
  Arms: Normal Saline

SUMMARY:
POEM (Peroral Endoscopic Myotomy) is an endoscopic procedure most commonly used to treat achalasia. Achalasia is a disorder resulting from the inability of esophageal muscles to relax.The POEM procedure, performed under general anesthesia, involves inserting an endoscope into the esophagus where a specialized knife is able to cut a new pathway through the esophageal tissue. The knife is then used to incise, and therefore loosen, tight muscles within the esophagus, lower esophageal sphincter, and the upper region of the stomach that are responsible for the symptoms.This study seeks to improve patient's post-operative pain levels by placing ropivacaine (a local anesthetic) into the newly cut pathway that is created in the POEM procedure. It is hypothesized that the topical irrigation of the POEM tunnel with ropivacaine will result in decreased pain scores and a decreased need for additional pain medications.

DETAILED DESCRIPTION:
POEM (Peroral Endoscopic Myotomy) is an endoscopic procedure most commonly used to treat achalasia. Achalasia is a disorder resulting from the inability of esophageal muscles to relax. Consequently, patients experience difficulty swallowing, reflux, and weight loss. Treatment options for achalasia are generally divided into 2 categories: A) treatment with medication, or B) treatment via a procedure. Medical treatment is generally reserved for patients to unwell to undergo procedures as the efficacy is low. Additionally, patients tend to experience many side-effects. There are also procedural options used to treat achalasia which include surgical myotomy and POEM. The POEM procedure is advantageous because it is less invasive, but is at least as equally effective for symptomatic relief when compared to the surgical myotomy. The POEM procedure, performed under general anesthesia, involves inserting an endoscope into the esophagus where a specialized knife is able to cut a new pathway through the esophageal tissue. The knife is then used to incise, and therefore loosen, tight muscles within the esophagus, lower esophageal sphincter, and the upper region of the stomach that are responsible for the symptoms. At the conclusion of the procedure, clips are placed in the esophagus to close the incision. Currently, patients are given intravenous ketorolac, oral viscous lidocaine and narcotic analgesics as needed to manage post-operative pain. This study, however, seeks to improve patient's post-operative pain levels by placing ropivacaine (a local anesthetic) into the newly cut pathway that is created in the POEM procedure. It is hypothesized that the topical irrigation of the POEM tunnel with ropivacaine will result in decreased pain scores and a decreased need for additional pain medications. Patients consented to participate in the study will be randomized to receive either ropivacaine (intervention group) or saline (control group). Pain will be assessed at 0.5, 1, 2, 4, and 6 hours post-admission to the recovery unit using validated pain scales. Additionally, the Quality of Recovery (QoR-15) patient survey, will be completed prior to discharge. This measure will capture the patient's initial post-operative health condition and help capture the overall patient experience.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older undergoing POEM procedure
* Able to provide written informed consent
* Fluent and literate in English

Exclusion Criteria:

* Patients with known adverse reactions to local anesthetics and NSAIDs (GFR<50)
* Patients with chronic pain taking regular analgesics or narcotics (requiring daily opioid therapy > 30 mg morphine or equivalents)
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Post-POEM pain level | 6 hours post-POEM procedure
  To assess the effect of the intervention/placebo on pain 6-hours post-POEM as assessed via the Numeric Rating Scale (NRS): The patient will be asked to rate their pain on a scale of 0-10, 0 representing no pain, and 10 representing the worst pain they have ever felt in their life.

SECONDARY OUTCOMES:
Post-POEM pain level | 0, 0.5, 1, 2, 4 hours post-POEM procedure
  Assessing pain scores at 0, 0.5, 1, 2, 4 hours post-POEM and on discharge
Quality of Recovery (QoR-15) score on the day of discharge | Assessed up to 24 hours post-POEM procedure
  Quality of Recovery-15 score: This survey captures patient's initial post-operative health condition and their overall patient experience. The patient will be asked to rate various emotional and physical aspects of their post-operative condition on a scale of 0-10. 0 will represent an emotion or activity experienced or accomplished none of the time, and 10 will represent an emotion or activity accomplished all of the time. Scores are summed; higher scores indicate a more optimal post-operative condition.
Post-POEM analgesic | 0 -6 hours post-procedure
  The requirement of post-POEM analgesic
Adverse Events | Assessed up to 24 hours post-POEM procedure
  Adverse events in hospital
Fentanyl consumption | Intra-procedure
  Intraprocedural fentanyl consumption
Repeatability of procedure | Assessed 24 hours post-POEM procedure
  Patient's willingness to have the procedure done on an outpatient basis: Patients will be asked if they are "willing" or "not willing" to have the procedure done on an outpatient basis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bechara, M.D., Principal Investigator — Queens University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadowski DC, Ackah F, Jiang B, Svenson LW. Achalasia: incidence, prevalence and survival. A population-based study. Neurogastroenterol Motil. 2010 Sep;22(9):e256-61. doi: 10.1111/j.1365-2982.2010.01511.x. Epub 2010 May 11. PMID 20465592
- [Background] Samo S, Carlson DA, Gregory DL, Gawel SH, Pandolfino JE, Kahrilas PJ. Incidence and Prevalence of Achalasia in Central Chicago, 2004-2014, Since the Widespread Use of High-Resolution Manometry. Clin Gastroenterol Hepatol. 2017 Mar;15(3):366-373. doi: 10.1016/j.cgh.2016.08.030. Epub 2016 Aug 28. PMID 27581064
- [Background] Goyal RK, Chaudhury A. Physiology of normal esophageal motility. J Clin Gastroenterol. 2008 May-Jun;42(5):610-9. doi: 10.1097/MCG.0b013e31816b444d. PMID 18364578
- [Background] Goyal RK, Chaudhury A. Pathogenesis of achalasia: lessons from mutant mice. Gastroenterology. 2010 Oct;139(4):1086-90. doi: 10.1053/j.gastro.2010.08.013. Epub 2010 Aug 25. No abstract available. PMID 20800108
- [Background] Clark SB, Rice TW, Tubbs RR, Richter JE, Goldblum JR. The nature of the myenteric infiltrate in achalasia: an immunohistochemical analysis. Am J Surg Pathol. 2000 Aug;24(8):1153-8. doi: 10.1097/00000478-200008000-00014. PMID 10935657
- [Background] Robertson CS, Martin BA, Atkinson M. Varicella-zoster virus DNA in the oesophageal myenteric plexus in achalasia. Gut. 1993 Mar;34(3):299-302. doi: 10.1136/gut.34.3.299. PMID 8386130
- [Background] Castagliuolo I, Brun P, Costantini M, Rizzetto C, Palu G, Costantino M, Baldan N, Zaninotto G. Esophageal achalasia: is the herpes simplex virus really innocent? J Gastrointest Surg. 2004 Jan;8(1):24-30; discussion 30. doi: 10.1016/j.gassur.2003.10.004. PMID 14746832
- [Background] Niwamoto H, Okamoto E, Fujimoto J, Takeuchi M, Furuyama J, Yamamoto Y. Are human herpes viruses or measles virus associated with esophageal achalasia? Dig Dis Sci. 1995 Apr;40(4):859-64. doi: 10.1007/BF02064992. PMID 7720482
- [Background] Birgisson S, Galinski MS, Goldblum JR, Rice TW, Richter JE. Achalasia is not associated with measles or known herpes and human papilloma viruses. Dig Dis Sci. 1997 Feb;42(2):300-6. doi: 10.1023/a:1018805600276. PMID 9052510
- [Background] Verne GN, Sallustio JE, Eaker EY. Anti-myenteric neuronal antibodies in patients with achalasia. A prospective study. Dig Dis Sci. 1997 Feb;42(2):307-13. doi: 10.1023/a:1018857617115. PMID 9052511
- [Background] Kallel-Sellami M, Karoui S, Romdhane H, Laadhar L, Serghini M, Boubaker J, Lahmar H, Filali A, Makni S. Circulating antimyenteric autoantibodies in Tunisian patients with idiopathic achalasia. Dis Esophagus. 2013 Nov-Dec;26(8):782-7. doi: 10.1111/j.1442-2050.2012.01398.x. Epub 2012 Sep 4. PMID 22947106
- [Background] Vaezi MF, Pandolfino JE, Vela MF. ACG clinical guideline: diagnosis and management of achalasia. Am J Gastroenterol. 2013 Aug;108(8):1238-49; quiz 1250. doi: 10.1038/ajg.2013.196. Epub 2013 Jul 23. PMID 23877351
- [Background] Schlottmann F, Herbella F, Allaix ME, Patti MG. Modern management of esophageal achalasia: From pathophysiology to treatment. Curr Probl Surg. 2018 Jan;55(1):10-37. doi: 10.1067/j.cpsurg.2018.01.001. Epub 2018 Jan 31. No abstract available. PMID 29548347
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] Schlottmann F, Luckett DJ, Fine J, Shaheen NJ, Patti MG. Laparoscopic Heller Myotomy Versus Peroral Endoscopic Myotomy (POEM) for Achalasia: A Systematic Review and Meta-analysis. Ann Surg. 2018 Mar;267(3):451-460. doi: 10.1097/SLA.0000000000002311. PMID 28549006
- [Background] Ujiki MB, Yetasook AK, Zapf M, Linn JG, Carbray JM, Denham W. Peroral endoscopic myotomy: A short-term comparison with the standard laparoscopic approach. Surgery. 2013 Oct;154(4):893-7; discussion 897-900. doi: 10.1016/j.surg.2013.04.042. PMID 24074429
- [Background] de La Coussaye JE, Eledjam JJ, Brugada J, Sassine A. [Cardiotoxicity of local anesthetics]. Cah Anesthesiol. 1993;41(6):589-98. French. PMID 8287299
- [Background] Scott DB, Lee A, Fagan D, Bowler GM, Bloomfield P, Lundh R. Acute toxicity of ropivacaine compared with that of bupivacaine. Anesth Analg. 1989 Nov;69(5):563-9. PMID 2679230